CLINICAL TRIAL: NCT06340165
Title: A Real-world Study of the Efficacy and Safety of Amlotinib for the Treatment of HER2-negative Advanced Breast Cancer
Brief Title: A Real-world Efficacy and Safety Study of Amlotinib for HER2-negative Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KS-151
Record Dates: First submitted 2024-01-01; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Anlotinib — Anrotinib is available in 12 mg, 10 mg, and 8 mg doses. The recommended dose of Anrotinib is 12 mg taken by mouth once daily, continuously, for 2 weeks on and 1 week off, in a 21-day cycle.

SUMMARY:
This study analyses the efficacy and safety of amlotinib as a study drug in the treatment of HER-2 negative advanced breast cancer in the real world, including the number of treatment lines, monotherapy, combination therapy, and different molecular subtypes of breast cancer. Evidence-based medicine evidence for clinicians. Although the clinical application of amlotinib in breast cancer treatment is a supra-indication drug, in view of its high safety and possible good efficacy for advanced breast cancer, some patients have been clinically adopted to try the treatment after communicating with their families. This study provides evidence for the further use of amlotinib in breast cancer treatment by analysing the efficacy and safety of amlotinib in real-world applications.

DETAILED DESCRIPTION:
The sample size was calculated according to the One-Sample Log-rank Test.During the treatment of amlotinib, metastatic site imaging was performed every 2-3 cycles, and the efficacy assessment and safety information were collected according to the RECIST version 1.1 criteria. After the completion of amlotinib treatment, survival follow-up was continued to clarify the survival status of the patients. When descriptive statistical analyses of clinicopathological characteristics were performed, categorical information was described by frequency counts and constitutive ratios, and quantitative information, such as conforming to normal distribution, was described by mean ± standard deviation, and not conforming to normal distribution, was described by median and interquartile spacing. Progression-free survival and overall survival at each time point were calculated by the Kaplan-Meier method and plotted as survival curves, Log-rank test was used to compare the prognostic differences between groups of latent variables, and the prognostic impact of latent variables on the anilotinib-treated patients was analysed using the COX regression risk model for exploratory analysis, and the risk ratios (hazard ratios (HRs) for quantitative evaluation. Variables with p-values less than 0.1 in the univariate COX regression analyses were screened by stepwise regression into the multivariate COX regression analyses. If the lapse rate exceeded 20%, sensitivity analyses were used to assess the impact of the lapse on the endpoint outcome event, which was performed by assuming a death outcome for the study subjects who were lost and analysing the endpoint event, and then treating the lost patients as normal and analysing the endpoint event and assessing the impact of the lost patients on the endpoint event. spss version 21.0 was used for the statistics, and a p<0.05 was considered to be clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* Imaging or tissue/cell puncture, etc. confirmed recurrent, metastatic breast cancer
* Pathologically confirmed HER-2 negative
* Application of amlotinib treatment until disease progression or toxicity intolerable, or voluntarily give up the continuation of amlotinib treatment,amlotinib application for at least 2 cycles
* The clinical data are basically complete

Exclusion criteria:

* Patients receiving local treatment means such as surgery and radiotherapy
* Patients with combined second primary breast cancer and other primary malignant tumors
* Patients with symptomatic brain metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective cohort study to collect clinical data of patients with HER-2 negative advanced breast cancer treated with amrutinib at four centers four centers at the First Hospital of Jilin University, Liaoning Provincial Cancer Hospital, Shandong Provincial Cancer Hospital, and Peking University Cancer Hospital between 2019.1 and 2022.9
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
PFS | Incorporation January 2021 through November 2023
  Progression-FreeSurvival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jilin University, Changchun, Jilin, China